CLINICAL TRIAL: NCT03820687
Title: Improving Informed Decision Making for Cancer Clinical Trial Participation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Patricia Chalela, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC20180283H
Record Dates: First submitted 2019-01-03; First posted 2019-01-29 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Participants in the intervention group will receive 3 components: 1) a bilingual, culturally tailored clinical trial educational video, 2) a low literacy booklet, and 3) support from a patient navigator to empower cancer patients to make informed decisions about cancer clinical trial participation by increasing awareness of clinical trials and MCC services, positive attitudes and intentions to consider clinical trials as an appropriate treatment option for cancer.
  Interventions: Other: Clinical Trial Educational Video; Other: Low literacy booklet; Other: Navigator
- Usual Care Control Group (Active Comparator): Participants in the usual care control group will receive a general clinical trial fact sheet.
  Interventions: Other: Clinical Trial Fact Sheet

INTERVENTIONS:
Other: Clinical Trial Educational Video — Bilingual, culturally tailored educational video, low literacy booklet, and support from a patient navigator to empower new cancer patients to make informed decisions about cancer clinical trial participation.
  Arms: Intervention Group
Other: Clinical Trial Fact Sheet — General Clinical Trial fact sheet with usual care information regarding Clinical Trials.
  Arms: Usual Care Control Group
Other: Low literacy booklet — A bilingual low-literacy booklet with educational content about clinical trials.
  Arms: Intervention Group
Other: Navigator — Support will be provided by a patient navigator to empower cancer patients to make an informed decision about cancer clinical trial participation by increasing awareness of clinical trials and MCC services, positive attitudes, and intentions to consider clinical trials as an appropriate treatment option for cancer.
  Arms: Intervention Group

SUMMARY:
The goal of this study is to develop and pilot test a multi-communication approach to improve informed decision-making about cancer Clinical Trials (CTs) participation by increasing awareness of CTs and Mays Cancer Center (MCC) services (treatment care capacities, reputation and resources), positive attitudes towards CTs, self-efficacy and intentions to consider CTs as an appropriate treatment option for cancer (intention to participate) among patients attending the MCC (clinic-based setting) and the general public in selected Bexar County areas (community-based settings).

DETAILED DESCRIPTION:
The proposed two-year study involves a randomized controlled educational trial featuring a 2-group parallel cohort design with random assignment of 400 cancer patients from the MCC to the intervention or usual care control group. Intervention participants will receive 3 components: 1) a bilingual culturally relevant educational video, 2) a low-literacy booklet and 3) support from a patient navigator to empower new cancer patients to make informed decisions about cancer CT participation by increasing awareness of clinical trials and MCC services, positive attitudes and intentions to consider CTs as an appropriate treatment option for cancer. The usual care control group will receive a general CT fact sheet.

The community setting will involve a community awareness campaign including 400 community members, with 3 components: 1) an educational session delivered via PowerPoint presentation or flip chart, 2) a low-literacy booklet, and 3) support from a community health educator to raise awareness, positive attitudes and intentions to consider CTs as an appropriate treatment option for cancer and promote the MCC services among community members in Bexar County.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cancer patients (within 1 year) attending any of the clinics at the MCC
* Patients who have not participated in a Clinical Trial before
* English or Spanish-speaking
* Able to provide informed consent

Exclusion Criteria:

* Younger than 18 years
* Patients who have already had a consultation with their doctor to discuss treatment options
* Patients who have participated in a Clinical Trial before
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who show intention to participate or to consider CTs as an appropriate treatment option for cancer. | Up to 3 months after the index oncology visit
  The percentage of patients who increased intentions to participate in a CT after the intervention compared with baseline.

SECONDARY OUTCOMES:
Proportion of patients who show increase in knowledge/awareness regarding CT participation. | Up to 3 months after the index oncology visit
  The percentage of patients who improved knowledge/awareness about clinical trials after the intervention compared with baseline.
Proportion of patients who show improved attitudes regarding CT participation. | Up to 3 months after the index oncology visit
  The percentage of patients who improve their attitudes towards clinical trial participation after the intervention compared with baseline.
Proportion of patients eligible for designated clinical trials who actually enroll in one of these trials. | Up to 3 months after the index oncology visit
  The percentage of patients who actually participate, or enroll in a clinical trial if they meet the eligibility criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Amelie G Ramirez, DrPH, MPH, Principal Investigator — UT Health San Antonio; Patricia Chalela, DrPH, MPH, Principal Investigator — UT Health San Antonio
Locations (1):
- University of Texas Health Science Center San Antonio, MCC, San Antonio, Texas, United States